CLINICAL TRIAL: NCT06302140
Title: A Phase 1 Study to Investigate the Mass Balance of [14C]-Nanatinostat and to Evaluate the Relative Bioavailability of Nanatinostat in Patients With Selected Advanced Cancers
Brief Title: A Mass Balance Study of [14C]-Nanatinostat and Relative Bioavailability Study of Nanatinostat in Patients With Advanced Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Viracta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VT3996-102
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Tablets; Valganciclovir

STUDY DESIGN:
Intervention Model Description: This clinical trial is divided into 3 parts (Part A, Part B, and Part C).
  Patients may begin their study participation in Part A or Part B. Part B (for patients who participate in Part A) and Part C (for patients who participate in Part A and/or Part B) are optional for patients who meet certain conditions for crossover.
  In Part A, patients will be given a single dose of radiolabeled nanatinostat by mouth on Day 1. Patients may stay in the hospital up to 8 days.
  In Part B, patients will receive both nanatinostat in a salt form and a non-salt form, coadministered with valganciclovir in different order across 2 treatment days. Patients will be randomly assigned to either receive the salt or the non-salt form of nanatinostat first. Patients may stay in the hospital up to 4 days.
  Part C will allow patients to continue receiving nanatinostat treatment as long as they are deriving clinical benefit. This part will not require a hospital stay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: [14C]-Nanatinostat (Experimental)
  Interventions: Drug: [14C]-Nanatinostat
- Part B (Treatment A): Nanatinostat (free base) tablets in combination with Valganciclovir (Experimental): Patients will be randomized into 2 treatment sequences (AB and BA) in Periods 1 and 2. Each treatment period is 24 hours.
  Interventions: Drug: Nanatinostat (free base) tablets in combination with Valganciclovir
- Part B (Treatment B): Nanatinostat mesylate tablets in combination with Valganciclovir (Experimental): Patients will be randomized into 2 treatment sequences (AB and BA) in Periods 1 and 2. Each treatment period is 24 hours.
  Interventions: Drug: Nanatinostat mesylate tablets in combination with Valganciclovir
- Part C: Single-agent Nanatinostat (free base) tablets (Experimental)
  Interventions: Drug: Single-agent Nanatinostat (free base) tablets

INTERVENTIONS:
Drug: [14C]-Nanatinostat — A single oral dose administered on Day 1 in a fasted state.
  Arms: Part A: [14C]-Nanatinostat
Drug: Nanatinostat (free base) tablets in combination with Valganciclovir — Treatment A: a single, oral dose of nanatinostat (free base) tablets (20 mg) in combination with valganciclovir (900 mg) under fed conditions.
  Arms: Part B (Treatment A): Nanatinostat (free base) tablets in combination with Valganciclovir
Drug: Nanatinostat mesylate tablets in combination with Valganciclovir — Treatment B: a single, oral dose of nanatinostat mesylate tablets (20 mg) in combination with valganciclovir (900 mg) under fed conditions.
  Arms: Part B (Treatment B): Nanatinostat mesylate tablets in combination with Valganciclovir
Drug: Single-agent Nanatinostat (free base) tablets — 40 mg once daily under fed conditions until disease progression or unacceptable toxicity, whichever occurs first.
  Arms: Part C: Single-agent Nanatinostat (free base) tablets

SUMMARY:
This study will determine how nanatinostat is absorbed, modified, and removed from the body (Part A), the amount of nanatinostat that becomes available to the body (Part B), and will evaluate the safety and tolerability of nanatinostat (Part C) in patients with advanced cancers.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, 3-part study evaluating the mass balance, pharmacokinetics, and metabolism of nanatinostat following a single oral dose of [14C]-nanatinostat for Part A, evaluating relative bioavailability of nanatinostat mesylate and nanatinostat (free base) tablets after coadministration with valganciclovir in patients with advanced stage cancers for Part B, and evaluating the safety and antitumor activity of nanatinostat for Part C.

The study was terminated prematurely and did not reach its target enrollment.

ELIGIBILITY:
Key Inclusion Criteria:

* Have histologically confirmed advanced stage cancers (excluding gastrointestinal tumors), have received standard therapies appropriate for their tumor type and stage with disease progression on or after the most recent treatment, and have no available treatment with curative intent.
* Eastern Cooperative Oncology Group Performance Status of ≤2 at Screening.
* Body mass index ≥18.5 but ≤30.0 kg/m2 at Screening.
* Adequate bone marrow, liver, and kidney function.

Key Exclusion Criteria:

* Presence of active central nervous system and/or leptomeningeal disease.
* Anticancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy, or use of other investigational agents within 4 weeks before study entry.
* Inability to take or tolerate oral medication.
* Any gastrointestinal, liver, or kidney condition that may affect drug absorption and metabolism.
* Active infection requiring systemic therapy.
* Has received radiolabeled material <12 months (excluding that required for imaging) prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
The amount of radioactivity in excreta [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: area under the plasma concentration versus time curve (AUC) [Part B] | 8 weeks after the last discharge visit in Part B
Pharmacokinetic Parameter: maximum plasma concentration (Cmax) [Part B] | 8 weeks after the last discharge visit in Part B
Pharmacokinetic Parameter: time to maximum observed plasma concentration (Tmax) [Part B] | 8 weeks after the last discharge visit in Part B
Pharmacokinetic Parameter: Fraction of the administered dose in comparison with a standard (Frel) [Part B] | 8 weeks after the last discharge visit in Part B
Incidence of adverse events and serious adverse events [Part C] | 28 days after the last dose of study treatment in Part C

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events [Parts A and B] | Up to 7 days after the last discharge visit
Incidence of clinically significant changes in selected safety assessments [Parts A and B] | Up to 7 days after the last discharge visit
Pharmacokinetic Parameter: area under the plasma concentration versus time curve (AUC) [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: maximum plasma concentration (Cmax) [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: time to maximum observed plasma concentration (Tmax) [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: elimination half-life (t1/2) [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: apparent total clearance (CL/F) [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: apparent volume of distribution during terminal phase (Vz/F) [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: elimination rate constant from the central compartment (Kel) [Part A] | 8 weeks after the last discharge visit in Part A
The ratio of total radioactivity in blood relative to plasma [Part A] | 8 weeks after the last discharge visit in Part A
[14C]-metabolic profile and identification of metabolites in plasma [Part A] | 8 weeks after the last discharge visit in Part A
Major radioactive peak/metabolites in urine and fecal radiochromatograms as a percentage of the radioactive dose [Part A] | 8 weeks after the last discharge visit in Part A
Pharmacokinetic Parameter: elimination half-life (t1/2) [Part B] | 8 weeks after the last discharge visit in Part B
Pharmacokinetic Parameter: metabolite-to-parent ratio [Part B] | 8 weeks after the last discharge visit in Part B
Objective Response Rate (ORR) [Part C] | Approximately 1 year
Time to Response (TTR) [Part C] | Approximately 1 year
Duration of Response (DOR) [Part C] | Approximately 1 year
Disease Control Rate (DCR) [Part C] | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Cohen, MD, PhD, Study Director — Viracta Therapeutics, Inc.
Locations (1):
- START Madrid - CIOCC - Hospital Universitario HM Sanchinarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No